CLINICAL TRIAL: NCT07196124
Title: Clinical Study Evaluating the Safety and Efficacy of BCMA/GPRC5D CAR-T in Patients With Relapsed/Refractory Multiple Myeloma.
Brief Title: BCMA/GPRC5D CAR-T Therapy for Multiple Myeloma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YD-005
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma Refractory
Keywords: CAR-T

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA/GPRC5D CAR-T cell injection (Experimental): Dose escalation: Three dose levels were designed, and if the maximum tolerated dose (MTD) was not found at the highest level, no further dose escalation was to be performed. Approximately 12-18 subjects were planned to be enrolled in the dose-escalation phase to evaluate the safety and tolerability of CAR-T injection and to determine the MTD and/or the recommended phase II dose (RP2D). Dose Expansion: During or after the dose escalation process, if a certain dose group is determined to have preliminary anti-tumor effects and controllable safety, it can be extended at this dose level to further evaluate the tolerance and safety of CAR-T injection, and to preliminarily evaluate its effectiveness.
  Interventions: Biological: BCMA/GPRC5D CAR-T

INTERVENTIONS:
Biological: BCMA/GPRC5D CAR-T — A single infusion of BCMA/GPRC5D CAR-T Injection administered intravenously.

SUMMARY:
This study is a single-arm, multicenter clinical trial of dose escalation and dose expansion.

DETAILED DESCRIPTION:
This study is a single-arm, mult-center clinical trial of dose escalation and dose expansion, primarily aimed at evaluating the safety, tolerability, and preliminary efficacy of BCMA/GPRC5D CAR-T cell infusion in subjects with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their guardian understands and voluntarily signs the informed consent form and expects to complete the follow-up examinations and treatments of the research protocol；
2. Age 18-85 years old (inclusive), gender unrestricted;
3. In accordance with the standards for the recurrence of multiple myeloma in the 'Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma (Revised 2022)';
4. Determine the presence of measurable lesions during screening based on any of the following criteria: serum monoclonal protein (M-protein) level ≥ 1.0 g/dL or urine M protein level ≥ 200 mg/24 hours; or diagnosed with light chain multiple myeloma without measurable lesions in serum or urine: serum immunoglobulin free light chain ≥ 10 mg/dL and serum immunoglobulin κ/γ free light chain ratio abnormal;
5. Has previously received at least first-line or higher treatment for multiple myeloma.
6. Patients with lymphoma must have at least one measurable lesion from baseline according to the revised IWG criteria for assessing the efficacy of malignant lymphoma；
7. The organ functions well；
8. ECOG performance status score 0-3 and estimated survival time greater than 3 months.

Exclusion Criteria:

1. Diagnosed with or treated for other invasive malignant tumors, excluding multiple myeloma, within 3 years;
2. Previous anti-tumor treatments (before the collection and preparation of CAR-T blood): received targeted therapy, epigenetic therapy, or experimental drug treatment within 14 days or within at least 5 half-lives (whichever is shorter), or used invasive experimental medical devices; received monoclonal antibody treatment for multiple myeloma within 21 days; received cytotoxic treatment within 14 days; received proteasome inhibitor treatment within 14 days; received immunomodulator treatment within 7 days; received radiotherapy within 14 days (except when the irradiated field covers ≤5% of the bone marrow reserve);
3. During screening, individuals with Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes), or primary AL amyloidosis;
4. Hepatitis B surface antigen (HBsAg) positive, hepatitis B core antibody (HBcAb) positive and peripheral blood HBV-DNA higher than the detection limit; Hepatitis C virus (HCV) antibody positive; Persons with human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA positive cases; EBV-DNA positive patients; The syphilis antibody was positive.
5. Those with a history of anaphylaxis [A history of anaphylaxis was defined as an allergic reaction of grade 2 or higher, in which any of the following clinical manifestations occurred: Airway obstruction (rhinorrhea, cough, stridor, dyspnea), Tachycardia, Hypotension, Arrhythmia, Gastrointestinal symptoms (nausea, vomiting), Incontinence, Laryngeal edema, Bronchospasm, Cyanosis, Shock, Respiratory, cardiac arrest] or known to be allergic to any of the drug active ingredients, excipents, or mouse-derived products or xenoproteins included in this trial (including the lymphatic cells clearance protocol).
6. Have severe cardiac disease, including but not limited to severe arrhythmia, unstable angina, massive myocardial infarction, New York Heart Association class III or IV cardiac dysfunction, and refractory hypertension.
7. Screen for patients who have had acute/chronic graft-versus-host disease (GVHD) within the past 6 months, or who require immunosuppressive treatment for GVHD;
8. Active autoimmune or inflammatory diseases (e.g., Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES)).
9. Patients with cancer emergencies (such as spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome, etc.) requiring emergency treatment before screening or reinfusion.
10. Presence of uncontrolled bacterial, fungal, viral, or other infection requiring antibiotic treatment.
11. Patients who had undergone major surgery (excluding diagnostic surgery and biopsy) within 4 weeks before lymphatic cells clearance or planned to undergo major surgery during the study period, or who had not fully healed the surgical wound before enrollment.
12. Persons with severe mental illness.
13. Within 1 week before the collection of peripheral blood mononuclear cells (PBMC), patients who use granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF) and other hematopoietic cytokine drugs that have an impact on the patient's blood picture (if it is a long-acting preparation, it is 2 weeks) and have an impact on cell preparation as judged by the investigator .
14. Within 2 weeks before PBMC collection, patients were receiving hormonal or immunosuppressive drugs that were judged by the investigator to have an effect on cell production.

    1. hormone: subjects who were receiving systemic steroid therapy within 2 weeks before PBMC collection and who required long-term systemic steroid therapy (except inhaled or topical use) as judged by the investigator during the treatment.
    2. Immunosuppressive agents: those who were receiving immunosuppressive agents within 2 weeks before PBMC collection.
15. Vaccination with live (attenuated) virus vaccine within 4 weeks prior to screening.
16. Alcoholics or those with a history of substance abuse.
17. Patients who, in the investigator's judgment and/or clinical criteria, have contraindications to any study procedure or other medical conditions that may put them at unacceptable risk.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2028-10-09 (Estimated); Study Completion 2028-12-09 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity Rate | Up to 28 days after CAR-T infusion.
  After the infusion of CAR-T, subjects still experienced adverse events, meeting the DLT definition, related to or possibly related to CAR-T infusion after optimal supportive treatment.
Incidence of Treatment-Emergent Adverse Events | Up to 24 months.
  Count the Incidence of adverse events.

SECONDARY OUTCOMES:
Concentration of CAR-T cells after Infusion (PK) | Up to 24 months.
  CAR-T in peripheral blood after infusion
Concentration of Cytokine after Infusion (PD) | Up to 24 months.
  Calculate the change of cytokine concentration in peripheral blood after After CAR-T infusion. Cytokines include IL-2、IL-6 and so on.
overall response rate, ORR | Up to 24 months.